CLINICAL TRIAL: NCT01709760
Title: A Prospective, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicentre, Phase III Study to Evaluate the Efficacy and Safety of ENIA11 in Combination With Methotrexate Versus Methotrexate Alone in Patients With Rheumatoid Arthritis
Brief Title: A Phase III Study to Evaluate the Efficacy and Safety of ENIA11 in Combination With Methotrexate Versus Methotrexate Alone in Patients With RA
Acronym: ENIA11
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mycenax Biotech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TSHEN1101
Record Dates: First submitted 2012-10-16; First posted 2012-10-18 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Rheumatoid Arthritis
Keywords: ENIA11; MTX; RA; TNF
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- methotrexate & ENIA11 (Experimental): ENIA11 25 mg, sc twice weekly
  Interventions: Drug: Methotrexate; Drug: ENIA11
- methotrexate & Placebo (Active Comparator): Placebo, sc twice weekly
  Interventions: Drug: Methotrexate; Drug: Placebo

INTERVENTIONS:
Drug: Methotrexate — Methotrexate 15-25 mg/week
Drug: ENIA11 — ENIA11 25 mg, sc twice weekly
  Other Names: TuNEX
  Arms: methotrexate & ENIA11
Drug: Placebo — Placebo, sc twice weekly
  Arms: methotrexate & Placebo

SUMMARY:
A Prospective, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicentre, Phase III Study to Evaluate the Efficacy and Safety of ENIA11 in Combination with Methotrexate versus Methotrexate Alone in Patients with Rheumatoid Arthritis

DETAILED DESCRIPTION:
The objectives of the study are to evaluate the efficacy and safety of ENIA11 in combination with methotrexate versus methotrexate alone in patients with rheumatoid arthritis.

This is a multi-center, double-blind, randomized, parallel-group, placebo-controlled study to evaluate the efficacy and safety of ENIA11 in combination with methotrexate versus methotrexate alone in patients with rheumatoid arthritis.

Subject participation duration: A total of 28 weeks, including: 2 weeks of screening, 24 weeks of treatment and 2 weeks of follow-up

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥ 20 years old;
2. Patient meet ACR criteria for rheumatoid arthritis over 6 month duration;
3. Patient with active disease at the time of screening as defined by six or more swollen joints and six or more tender joints;
4. Presence of at least one of the following criteria:

   * Erythrocyte Sedimentation Rate (ESR) ≥ 28 mm/h,
   * C-Reactive Protein (CRP) ≥ 10 mg/L,
5. RA functional class I, II, or III;
6. Patients have been treated on methotrexate for at least 3 month, and maintained at stable dose of 15-25 mg/week for at least 8 weeks; MTX low dose as 10 mg per week is allowed for patients who had a documented history of constitutional symptoms at higher doses.
7. Patient is willing and able to comply with study procedures and sign informed consent.

Exclusion Criteria:

1. Active autoimmune disease (other than RA) requiring immunosuppressive therapy;
2. In the opinion of the investigator, the patient shows persistent signs of immunosuppression;
3. Known hypersensitivity to etanercept or ENIA11 or any of its components;
4. Previous unsuccessful treatment with etanercept, anti-TNF monoclonal antibodies or a soluble TNF receptor (e.g., infliximab);
5. Suspected or diagnosed pulmonary tuberculosis, or other chronic or current infectious disease at discretion of investigator;
6. Patients who have a history or evidence of a medical condition that would expose them to an undue risk of a significant adverse event during the course of the trial, including but not limited to hepatic, renal, respiratory, cardiovascular, endocrine, immune, neurological, hematological, gastrointestinal or psychiatric disease as determined by the clinical judgment of the investigator;
7. Patients with any of the following laboratory abnormalities: ALT/AST > 3 times ULN, creatinine > 2 mg/dl, WBC < 3,000/mm3, Hgb < 8.5 g/dL, platelet count < 100,000/mm3;
8. Patients have received live attenuated vaccination program within 3 months or BCG vaccine within 12 months prior enrollment;
9. Female patient of childbearing potential who:

   * is lactating; or
   * has positive urine pregnancy test at Visit 1; or
   * refuse to adopt reliable method of contraception during the study;
10. Diagnosis of primary fibromyalgia or other joint inflammatory disease including but not limited to gout, reactive arthritis, psoriatic arthritis, seronegative spondyloarthropathy, Lyme disease;
11. Known or suspected positive serology for human immunodeficiency, hepatitis B or C virus;
12. Patient has received any investigational agent within 28 days or 5 half-lives, whichever is longer, prior to the first dose of investigational product;
13. Patient has history of substance abuse, drug addiction or alcoholism;
14. Patient who have had participated in prior phase I/II clinical trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2012-11; Primary Completion 2017-12 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
ACR20 responder at last treatment visit | Week 24
  The primary efficacy endpoint is defined as ACR20 responder at last treatment visit (Week 24).

CONTACTS AND LOCATIONS:
Overall Officials: Joung-Liang Lan, PHD, Principal Investigator — China Medical University Hospital; Chung-Ming Huang, MD, Principal Investigator — China Medical University Hospital; Der-Yuan Chen, PHD, Principal Investigator — Taichung Veterans General Hospital; Ling-Ying Lu, PHD, Principal Investigator — Kaohsiung Veterans General Hospital.; Ning-Sheng Lai, PHD, Principal Investigator — Buddhist Tzu Chi General Hospital; Tien-Tsai Cheng, MD, Principal Investigator — Chang Gung Memorial Hospital; Gregory J Tsay, PHD, Principal Investigator — Chung Shan Medical University; Ying-Ming Chiu, MD, Principal Investigator — Changhua Christian Hospital
Locations (8):
- Taiwan (8):
  - Changhua Christian Hospital, Changhua
  - Buddhist Tzu Chi General Hospital, Chiayi City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - China Medical University Hospital, Taichung
  - Chung Shan Medical University Hospital, Taichung
  - Taipei City Hospital, Taipei